CLINICAL TRIAL: NCT00182780
Title: The Use of American Ginseng (Panax Quinquefolius) to Improve Cancer-Related Fatigue: A Randomized, Double-Blind, Dose-Finding, Placebo-Controlled Study
Brief Title: American Ginseng in Treating Patients With Cancer-Related Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NCCTG-N03CA; NCI-2012-02670 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000440907 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2005-09-15; First posted 2005-09-16 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Fatigue; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: fatigue; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Fatigue | interventions — Asian ginseng

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm I - American ginseng (low dose) (Experimental): Patients receive oral American ginseng twice daily for 8 weeks in the absence of unacceptable toxicity.
  After 8 weeks of treatment, patients in arms I-III may continue to receive American ginseng on the optional continuation portion of the study for an additional 8 weeks. Patients in arm IV may begin oral American ginseng twice daily for 8 weeks on the optional continuation portion of the study.
  Quality of life is assessed at baseline, every 2 weeks during treatment, and at the end of treatment.
  PROJECTED ACCRUAL: A total of 280 patients (70 per treatment arm) will be accrued for this study within 35 months.
  Interventions: Dietary Supplement: American ginseng
- Arm II - American ginseng (mid-dose) (Experimental): Patients receive oral American ginseng at the mid-dose twice daily for 8 weeks in the absence of unacceptable toxicity.
  After 8 weeks of treatment, patients in arms I-III may continue to receive American ginseng on the optional continuation portion of the study for an additional 8 weeks. Patients in arm IV may begin oral American ginseng twice daily for 8 weeks on the optional continuation portion of the study.
  Interventions: Dietary Supplement: American ginseng
- Arm III - American ginseng (high-dose) (Experimental): Patients receive oral American ginseng at the high dose twice daily for 8 weeks in the absence of unacceptable toxicity.
  After 8 weeks of treatment, patients in arms I-III may continue to receive American ginseng on the optional continuation portion of the study for an additional 8 weeks. Patients in arm IV may begin oral American ginseng twice daily for 8 weeks on the optional continuation portion of the study.
  Interventions: Dietary Supplement: American ginseng
- Arm IV - Placebo (Other): Patients receive oral placebo twice daily for 8 weeks in the absence of unacceptable toxicity.
  After 8 weeks of treatment, patients in arms I-III may continue to receive American ginseng on the optional continuation portion of the study for an additional 8 weeks. Patients in arm IV may begin oral American ginseng twice daily for 8 weeks on the optional continuation portion of the study.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: American ginseng
  Arms: Arm I - American ginseng (low dose); Arm II - American ginseng (mid-dose); Arm III - American ginseng (high-dose)
Other: Placebo
  Arms: Arm IV - Placebo

SUMMARY:
RATIONALE: American ginseng may help relieve cancer-related fatigue.

PURPOSE: This clinical trial is studying how well American ginseng works in treating patients with cancer-related fatigue.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the efficacy of American ginseng, administered at 3 different doses, vs placebo in patients with cancer-related fatigue.

Secondary

* Determine the toxic effects and tolerability of American ginseng in these patients.
* Determine the impact of American ginseng on quality of life-related variables (e.g., sleep, vitality, and quality of life domains) in these patients.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to disease stage (I or II vs III or IV vs unknown), gender (male vs female), baseline fatigue score (4-7 vs 8-10), concurrent chemotherapy (yes vs no), and concurrent radiotherapy (yes vs no). Patients are randomized to 1 of 4 treatment arms.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed cancer
* Experiences cancer-related fatigue, defined as a baseline fatigue score of ≥ 4 on a numerical analogue scale (0-10)

  * Fatigue must be present for ≥ 1 month before study entry
* No primary brain cancer, brain metastases, or other CNS malignancy, including CNS lymphoma

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* At least 6 months

Hematopoietic

* Hemoglobin ≥ 11 g/dL

Hepatic

* SGOT ≤ 1.5 times upper limit of normal (ULN)

Renal

* Calcium ≤ 1.2 times ULN
* Creatinine ≤ 1.2 times ULN

Cardiovascular

* No uncontrolled hypertension (i.e., diastolic blood pressure [BP] > 100 mm Hg and/or systolic BP > 160)

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No diabetes, defined as receiving oral hypoglycemics or insulin
* No hypersensitivity to ginseng
* No uncontrolled pain, hypothyroidism, or insomnia that is considered to be the primary cause of patient's fatigue
* Not currently under the care of a psychiatrist for documented psychiatric disorder (e.g., severe depression, manic depressive disorder, obsessive-compulsive disorder, or schizophrenia)

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Concurrent epoetin alfa for treatment of anemia allowed

Chemotherapy

* Concurrent chemotherapy allowed except CHOP therapy

Endocrine therapy

* No concurrent chronic systemic steroids

Radiotherapy

* Not specified

Surgery

* More than 4 weeks since prior major surgery

Other

* No prior ginseng capsules for fatigue

  * Prior ginseng-containing teas or drinks purchased at a grocery store allowed
* No concurrent pharmacologic agents for the treatment of fatigue, including any of the following:

  * Psychostimulants
  * Antidepressants

    * Antidepressants used to treat conditions other than fatigue (e.g., hot flashes) are allowed provided the patient has been on a stable dose for ≥ 1 month and plans to continue antidepressant for ≥ 1 month
* No concurrent monoamine oxidase inhibitors
* No concurrent full anticoagulation doses of warfarin or heparin

  * A dose of 1 mg/day for preventing catheter clots allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2005-10; Primary Completion 2006-09-05 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Fatigue by brief inventory at 4 and 8 weeks of treatment | at 4 and 8 weeks

SECONDARY OUTCOMES:
Sleep by Pittsburg Sleep Quality Inventory at 4 and 8 weeks of treatment | at 4 and 8 weeks
Quality of life by North Central Cancer Treatment Group Uniscale at 4 and 8 weeks of treatment | at 4 and 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Brent A. Bauer, MD, Study Chair — Mayo Clinic

REFERENCES:
- [Result] Barton DL, Soori GS, Bauer BA, Sloan JA, Johnson PA, Figueras C, Duane S, Mattar B, Liu H, Atherton PJ, Christensen B, Loprinzi CL. Pilot study of Panax quinquefolius (American ginseng) to improve cancer-related fatigue: a randomized, double-blind, dose-finding evaluation: NCCTG trial N03CA. Support Care Cancer. 2010 Feb;18(2):179-87. doi: 10.1007/s00520-009-0642-2. Epub 2009 May 6. PMID 19415341